CLINICAL TRIAL: NCT00385827
Title: A Phase 2, Multicenter, Open-Label Study of CNTO 328 (Anti-IL-6 Monoclonal Antibody) in Combination With Mitoxantrone Versus Mitoxantrone in Subjects With Metastatic Hormone-Refractory Prostate Cancer (HRPC)
Brief Title: A Safety and Efficacy Study of Siltuximab (CNTO 328) in Male Subjects With Metastatic Hormone-Refractory Prostate Cancer (HRPC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely stopped after Independent Data Monitoring Committee (IDMC) evaluation for lack of efficacy.
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012346; C0328T07; 2006-001671-38 (EudraCT Number)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Cancer, Prostate
Keywords: Cancer; Prostate; IL-6; Mitoxantrone; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Mitoxantrone; siltuximab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mitoxantrone+Prednisone+Siltuximab (CNTO 328) (Part 1) (Experimental): In Part 1, mitoxantrone 12 milligram per square meter (mg/m^2) will be given intravenously as a 30-minute infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with siltuximab 6 mg/kilogram (mg/kg) intravenously as a 2 hour-infusion every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year; and prednisone 5 mg orally twice daily starting with the first administration of mitoxantrone.
  Interventions: Drug: Mitoxantrone; Drug: Siltuximab; Drug: Prednisone
- Mitoxantrone+Prednisone+Siltuximab (Part 2) (Experimental): In Part 2, mitoxantrone 12 mg/m^2 will be given intravenously as a 30-minute infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with siltuximab 6 mg/kg intravenously as a 2-hour infusion every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year; and prednisone 5 mg orally twice daily starting with the first administration of mitoxantrone.
  Interventions: Drug: Mitoxantrone; Drug: Siltuximab; Drug: Prednisone
- Mitoxantrone+Prednisone (Part 2) (Active Comparator): In Part 2, mitoxantrone 12 mg/m^2 will be given intravenously as a 30-minute infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with prednisone 5 mg orally twice daily starting with the first administration of mitoxantrone.
  Interventions: Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Drug: Mitoxantrone — Mitoxantrone 12 mg/m^2 intravenously as a 30 minute infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2)
Drug: Siltuximab — Siltuximab 6 mg/kg intravenously as a 2 hour infusion every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year
  Other Names: CNTO 328
  Arms: Mitoxantrone+Prednisone+Siltuximab (CNTO 328) (Part 1); Mitoxantrone+Prednisone+Siltuximab (Part 2)
Drug: Prednisone — Prednisone 5 mg orally twice daily

SUMMARY:
The purpose of this study is to assess the safety and efficacy of siltuximab administered in combination with mitoxantrone and prednisone in participants with metastatic (spread of cancer cells from one part of the body to another) hormone-refractory (not responding to treatment) prostate cancer (abnormal tissue that grows and spreads in the body) (HRPC).

DETAILED DESCRIPTION:
This is a 2-part, open-label (all people know the identity of the intervention) multicenter (when more than 1 hospital or medical school team work on a medical research study), Phase 2 study to evaluate the safety and efficacy of the combination of siltuximab plus mitoxantrone versus mitoxantrone in participants with metastatic HRPC who have received 1 prior Docetaxel-based chemotherapy (treatment of disease, usually cancer, by chemical agents) regimen (pattern of giving treatment). Part 1 of the study is single arm where participants will receive mitoxantrone, prednisone and siltuximab. Part 2 of the study is randomized portion (the study drug is assigned by chance), consisting of 2-arms. The experimental arm will consist of treatment with mitoxantrone, prednisone and siltuximab. The control arm will consist of treatment with mitoxantrone and prednisone. Mitoxantrone will be administered at a dose of 12 milligram per square meter (mg/m^2) intravenously (into a vein) as a 30-minute infusion (a fluid or a medicine delivered into a vein by way of a needle) on Day 1 of each 3-week cycle, until disease progression or unacceptable toxicity (any harmful effect of a drug) or up to 10 cycles (a maximum total dose of approximately 120 mg/m^2). Siltuximab will be administered at a dose of 6 mg/kilogram intravenously as a 2-hour infusion, starting Day 1 of Cycle 1 to continue every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year. All participants will receive prednisone 5 mg twice daily starting with the first administration of Mitoxantrone. The duration of treatment will be a maximum of 12 months for cumulative dose. Radiologic assessments will be performed on Week 12 after the first study agent dosing, then every 9 weeks until the end of treatment and then once every 3 months until documented disease progression. Tumor (a mass in a specific area) response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. There will be short-term follow-up visits (conducted monthly for 2 months), followed by long-term follow-up visits (conducted once every 3 months). Participants' safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (the study of tissue under the microscope) or cytologically (the study of cells) confirmed adenocarcinoma (a malignant epithelial tumor with a glandular organization) of the prostate
* Radiologically (Gamma and Computed Topography [CT] scans) documented metastatic disease
* At least 6 weeks of treatment with 1 prior docetaxel-based chemotherapy for metastatic Hormone Refractory Prostate Cancer (HRPC)
* Disease progression, during or within 6 months of stopping of prior docetaxel-based therapy, based on one of the following: serum Prostate Specific Antigen (PSA) progression, defined as a rise in at least 2 consecutive serum PSA values, each obtained at least 1 week apart or radiologic disease progression: if disease progression is shown by bone scan only, then disease progression is defined by the appearance of 2 or more new bone lesions (abnormal area of tissue, such as a wound, sore, rash, or boil)
* Orchiectomy (surgery to remove one or both testicles) or testosterone less than 50 nanogram per decilliter (ng/dL) by means of pharmacological/chemical castration

Exclusion Criteria:

* No evidence of a brain tumor
* No more than 1 line of chemotherapy for metastatic prostate cancer
* No prior mitoxantrone treatment
* Prior malignancy (other than prostate cancer) except adequately treated superficial bladder cancer, basal cell or squamous cell carcinoma (type of cancer) of the skin, or other cancer for which the subject has been disease-free for atleast 3 years
* No Human Immunodeficiency Virus (HIV) (a life-threatening infection that you can get from an infected person's blood or from having sex with an infected person) seropositivity or hepatitis (inflammation of the liver) B or C infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (34):
- United States (11):
  - Norwalk, Connecticut
  - Port Saint Lucie, Florida
  - Atlanta, Georgia
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - St Louis, Missouri
  - New York, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - North Charleston, South Carolina
  - Milwaukee, Wisconsin
- Austria (4):
  - Innsbruck
  - Sankt Veit an der Glan
  - Vienna
  - Wels
- Belgium (7):
  - Aalst
  - Antwerp
  - Brasschaat
  - Brussels
  - Roeselare
  - Sint-Niklaas
  - Wilrijk
- France (4):
  - Caen
  - Le Mans
  - Lyon
  - Villejuif
- Germany (3):
  - Berlin
  - Cologne
  - Kassel
- Spain (3):
  - Barcelona
  - Madrid
  - Málaga
- United Kingdom (2):
  - London
  - Sutton

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Mitoxantrone + Prednisone + Siltuximab: Participants received mitoxantrone 12 milligram per square meter (mg/m^2) intravenously (into a vein) as a 30-minute infusion (a fluid or a medicine delivered into a vein by way of a needle) on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with siltuximab (CNTO 328) 6 milligram per kilogram (mg/kg) intravenously as a 2-hour infusion every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year; and prednisone 5 milligram (mg) orally twice daily starting with the first administration of mitoxantrone.
- Part 2: Mitoxantrone + Prednisone: Participants received mitoxantrone 12 mg/m^2 intravenously as a 30-minute on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with prednisone 5 mg orally twice daily starting with the first administration of mitoxantrone.
- Part 2: Mitoxantrone + Prednisone + Siltuximab: Participants received mitoxantrone 12 mg/m^2 intravenously as a 30-minute infusion on Day 1 of each 3-week cycle until disease progression or unacceptable toxicity or up to 10 cycles (a maximum cumulative dose of approximately 120 mg/m^2) along with siltuximab 6 mg/kg intravenously as a 2-hour infusion every 2 weeks until disease progression or unacceptable toxicity or up to a maximum of 1 year; and prednisone 5 mg orally twice daily starting with the first administration of mitoxantrone.
Period: Part 1
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Started | 9 | 0 | 0
Treated | 9 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 9 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Started | 0 | 49 | 48
Treated | 0 | 47 | 46
Completed | 0 | 16 | 0
Not Completed | 0 | 33 | 48
Not completed — Adverse Event | 0 | 6 | 10
Not completed — Death | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 14 | 13
Not completed — Randomized but not treated | 0 | 2 | 2
Not completed — Other | 0 | 11 | 21

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who received at least one dose of study drug in Part 1 and all randomized participants in Part 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab | Total
Number analyzed (Participants) | 9 | 49 | 48 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.89) | 67.8 (7.83) | 67.9 (9.28) | 68 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 49 | 48 | 106
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 0 | 1 | 2 | 3
  BELGIUM | 0 | 6 | 6 | 12
  FRANCE | 0 | 15 | 12 | 27
  GERMANY | 0 | 4 | 5 | 9
  SPAIN | 0 | 7 | 4 | 11
  UNITED KINGDOM | 0 | 5 | 6 | 11
  UNITED STATES | 9 | 11 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Baseline up to 12 weeks after last dose administration
Population: Safety population in Part 1 included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 9
participants
  AEs | 9
  SAEs | 5

2. Primary Outcome: Part 2: Progression Free Survival (PFS)
Description: The PFS is the time from the date of randomization until the first documented sign of progression (at least a 20 percent increase in the sum of the longest diameter [LD] of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new target or non-target lesions as per Response Evaluation Criteria in Solid Tumors [RECIST] or 3 or more new skeletal lesions on bone scan with confirmation of second bone scan or with clinical deterioration) or death, whichever occurs first.
Time Frame: Randomization, Week 12, then every 9 weeks until 1 month after last dose administration, then every 3 months until disease progression or death, up to 2 years
Population: Intent-to-treat (ITT) population in Part 2 included all randomized participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 49 | 48
days | 228.0 [155.0 to 303.0] | 97.0 [84.0 to 179.0]

3. Secondary Outcome: Time to Clinical Deterioration (TtCD)
Description: The TtCD is defined as the time from the start of treatment (for participants in Part 1) or randomization (for participants in Part 2) until the first documented clinical deterioration (consists of pain requiring palliative (intended to relieve pain) intervention (a treatment given during the course of a research study), or death due to any cause, whichever occurs earlier.
Time Frame: Start of treatment (Part 1)/Randomization (Part 2), Week 1 of each cycle up to 1 month after last dose administration, and thereafter every 3 months until clinical deterioration or death, up to 2 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 9 | 49 | 48
days | 199.0 [107.0 to NA] — Upper limit of the confidence interval was not reachable as data was not matured at the time of the analysis, due to early study termination. | 298.0 [128.0 to 342.0] | 183.0 [142.0 to 274.0]

4. Secondary Outcome: Number of Participants With Palliative Response
Description: Palliative response was defined as a 2-point or greater reduction from baseline pain, without a categorical increase in prescribed disease-related analgesic (drug used to control pain) use or at least a categorical decrease in disease-related analgesic use without a concomitant (given at the same time) increase in pain. Each component required confirmation at least 3 weeks later.
Time Frame: Start of treatment (Part 1)/Randomization (Part 2), Week 1 of each cycle up to 1 month after last dose administration, and thereafter every 3 months up to 2 years
Population: Data for this outcome measure was not analyzed because minimal efficacy analysis (primary and key secondary endpoints) was done due to early termination of study.
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Prostate Specific Antigen (PSA) Response
Description: The PSA response is defined as at least a 50% reduction in PSA from the Baseline value, confirmed by a second PSA value at least 3 weeks after initial documentation of PSA response.
Time Frame: Start of treatment (Part 1)/Randomization (Part 2), Week 1 of each cycle up to 1 month after last dose administration, and thereafter every 3 months until disease progression, up to 2 years
Population: Analysis population included all participants who received at least one dose of study drug in Part 1 and all randomized participants in Part 2. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 9 | 46 | 45
participants | 4 | 12 | 7

6. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the date of start of treatment (for participants in Part 1) or randomization (for participants in Part 2) to death due to any cause. For participants who were alive at the time of analysis, OS was censored at the last contact date.
Time Frame: Start of treatment (Part 1)/Randomization (Part 2) until death, up to 2 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Number analyzed (Participants) | 9 | 49 | 48
days | 368.0 [214.0 to NA] — Upper limit of the confidence interval was not reachable as data was not matured at the time of the analysis, due to early study termination. | 394.0 [311.0 to 438.0] | 311.0 [226.0 to NA] — Upper limit of the confidence interval was not reachable as data was not matured at the time of the analysis, due to early study termination.

ADVERSE EVENTS:
Time Frame: Baseline up to 12 weeks after last dose administration
Description: Safety population in Part 1 and 2 included all participants who received at least one dose of study drug.
Arm/Group | Part 1: Mitoxantrone + Prednisone + Siltuximab | Part 2: Mitoxantrone + Prednisone | Part 2: Mitoxantrone + Prednisone + Siltuximab
Serious Adverse Events (participants affected / at risk) | 5/9 | 18/47 | 18/46
Other Adverse Events (participants affected / at risk) | 9/9 | 42/47 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Mitoxantrone + Prednisone + Siltuximab (N=9) | Part 2: Mitoxantrone + Prednisone (N=47) | Part 2: Mitoxantrone + Prednisone + Siltuximab (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Catheter Site Haemorrhage (General disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1
Disease Progression (General disorders) | 2 | 3 | 6
Fatigue (General disorders) | 1 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibrinolysis (Investigations) | 0 | 1 | 0
Fibrinolysis Increased (Investigations) | 0 | 0 | 1
International Normalised Ratio Decreased (Investigations) | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Facial Palsy (Nervous system disorders) | 0 | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 3
Venous Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Mitoxantrone + Prednisone + Siltuximab (N=9) | Part 2: Mitoxantrone + Prednisone (N=47) | Part 2: Mitoxantrone + Prednisone + Siltuximab (N=46)
Anaemia (Blood and lymphatic system disorders) | 6 | 11 | 4
Leukopenia (Blood and lymphatic system disorders) | 7 | 2 | 10
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 9 | 14 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3 | 11
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 3 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 4
Blindness (Eye disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 2
Visual Impairment (Eye disorders) | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 4 | 2
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 17 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 11
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 7 | 18
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2 | 6
Asthenia (General disorders) | 1 | 9 | 12
Chest Pain (General disorders) | 1 | 0 | 4
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 10 | 14
Oedema Peripheral (General disorders) | 1 | 0 | 5
Temperature Intolerance (General disorders) | 1 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Localised Infection (Infections and infestations) | 2 | 1 | 3
Rhinitis (Infections and infestations) | 3 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 2 | 3
International Normalised Ratio Increased (Investigations) | 1 | 0 | 0
Low Density Lipoprotein Increased (Investigations) | 1 | 0 | 0
Weight Decreased (Investigations) | 3 | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 4 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Enzyme Abnormality (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 7
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 6
Cerebral Ischaemia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 3
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 2 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 3 | 1
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 8
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 3
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1 | 4
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 3 | 3 | 0

LIMITATIONS AND CAVEATS:
Results of few secondary endpoints were not reported as the study was terminated early due to the premature suspension and subsequent halting of study enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less